CLINICAL TRIAL: NCT05812248
Title: Prediction of Vascular Events After Major Non-Cardiac Surgery : an Observational Prospective Cohort Study
Acronym: PREVENGE-CB-2
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-223
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Noncardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Perioperative cardiac biomarker measurement — High-sensitivity cardiac troponin T is measured within 7 days prior to surgery and at day 1 and day 2 after surgery. N-terminal pro-B-type natriuretic peptide is measured within 7 days before surgery.

SUMMARY:
This observational study includes patients at medium-to-high cardiovascular risks undergoing major noncardiac surgery, measures their baseline demographic and clinical characteristics, preoperative cardiac biomarkers and intraoperative surgery/anesthesia related data, and screens them for the occurrence of myocardial injury and major adverse cardiac events after surgery. The primary aim is to develop and validate a pre- and an immediate postoperative prediction model for occurrence of major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years;
* Undergoing major noncardiac surgery (expected procedure duration ≥2 h, expected length of postoperative stay ≥2 d);
* History of at least one cardiovascular disease (i.e., coronary artery disease, stroke, congestive heart failure, or peripheral arterial disease) or with at least two cardiovascular risk factors (i.e., hypertension, diabetes, chronic kidney disease, smoking in the past ≥2 years, ≥65 years of age, hypercholesterolemia, history of TIA, high-risk surgery (intrathoracic, intraperitoneal, or major vascular)).

Exclusion Criteria:

* History of acute cardiovascular events within 30 days prior to surgery;
* American Society of Anesthesiologists (ASA) physical status of 5 or greater;
* Previously enrolled in this study;
* Unable to understand or to sign informed consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major noncardiac suregry with medium-to-high risks for postoperative cardiac complications.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major adverse cardiac event | Within 30 days after the index surgery
  A composite outcome that includes cardiac death, myocardial infarction, non-fatal cardiac arrest, and coronary revascularisation.

SECONDARY OUTCOMES:
Number of patients with myocardial injury after noncardiac suregry (MINS) | Within 30 days after the index surgery
  MINS is defined as a postoperative hsTnT level of 20 to less than 65 ng/L with an absolute change of at least 5 ng/L or a postoperative hsTnT level of at least 65 ng/L. A 20% or greater increase of hsTnT level from preoperative baseline is required to exclude chronic troponin elevation. Troponin elevations believed to be consequent to nonischemic causes are excluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China